CLINICAL TRIAL: NCT06951542
Title: Improving HIV and Depression Outcomes by Reducing HIV-Mental Illness Stigma in Salima and Mulanje Districts: Pilot Trial
Brief Title: HIV-Mental Illness Stigma Reduction and Outcomes in Malawi
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melissa Stockton, Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 857336; 7K01MH130226-03 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-04-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; HIV; Health Condition Stigma
Keywords: Malawi; Health Condition Stigma; Stigma; Measurement-based Care (MBC); Friendship Bench (FB) Therapy; Salima; Mulanje; Mental Illness Stigma; HIV Stigma; Stigma Reduction Counseling; Stigma Intervention; Multi-Level Stigma Reduction; HIV Care Engagement; HIV; Depression
MeSH Terms: conditions — Social Stigma; Depression

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a pilot trial, with a multiple baseline design to enroll 200 depressed PLHIV at the study sites who will either receive usual depression care during the pre-implementation phase or enhance usual depression care (+ stigma-reduction counseling) during the implementation phase. Using the multiple baseline design with two phases (a pre-implementation phase and an intervention implementation phase), the intervention launches earlier at Clinic A than Clinic B, based on random selection. Staggering the launch of the implementation phase will allow for assessment of and potential correction for any secular trend in outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation Phase (No Intervention): In the pre-implementation phase, antiretroviral therapy (ART) providers will screen and treat patients at ART for depression as is now standard practice. Namely, patients will be screened using the Patient Health Questionnaire-9 (PHQ-9) and depressed patients will be treated with Measurement-based Care (MBC) and/or Friendship Bench (FB) problem-solving therapy. At each monthly ART appointment, providers assess patients' depressive symptoms and continue depression treatment as clinically indicated.
- Intervention Implementation Phase (Experimental): In the intervention implementation phase, patients at antiretroviral therapy (ART) will be screened and treated for depression as described and assessed for the study enrollment as in the pre-implementation phase. Depressed patients will be referred to counselors to receive the stigma-reduction intervention sessions. Stigma-reduction counseling sessions will include psychoeducation and activities to challenge myths and stereotypes, cope with experiences of discrimination, and overcome self-stigma. Intervention sessions will be audio-recorded (with participants' consent) as part of the fidelity assessment.
  Interventions: Behavioral: Stigma Reduction Counseling

INTERVENTIONS:
Behavioral: Stigma Reduction Counseling — The stigma reduction counseling sessions will include psychoeducation and activities to challenge myths and stereotypes, cope with experiences of discrimination, and overcome self-stigma.
  Arms: Intervention Implementation Phase

SUMMARY:
The overall aim of this study is to assess the acceptability, feasibility, fidelity, and effectiveness of a depression treatment intervention augmented with counseling to address stigma. Using a multiple-baseline design, 200 depressed adults living with HIV will be enrolled in the trial. Participant surveys and abstracted clinical data related to HIV and depression care will assess the effectiveness of the intervention.

DETAILED DESCRIPTION:
Stigma and depression are associated with increased HIV-related mortality and morbidity; as depression treatment is increasingly integrated into HIV care, addressing HIV stigma, mental illness stigma, and intersectional HIV-mental illness stigma is crucial. The Malawi Ministry of Health has recently integrated depression screening and treatment into the antiretroviral therapy (ART) departments of 12 District Hospitals across the country, including Salima and Mulanje District Hospital. Through this program, adults living with HIV are now screened with the Patient Health Questionnaire-9 (PHQ-9) and depressed patients are prescribed antidepressants using Measurement-based Care (MBC) or referred for Friendship Bench (FB) problem-solving therapy.

With this study the investigators aim to augment the existing depression treatment program at Salima and Mulanje District Hospitals with counselling to help address and reduce stigma. The stigma reduction counseling sessions will include psychoeducation and activities to challenge myths and stereotypes, cope with experiences of discrimination, and overcome self-stigma. Ultimately, this study will evaluate the feasibility, acceptability, fidelity, and preliminary effectiveness of the HIV-mental illness stigma-reduction intervention as part of depression treatment integrated into HIV care at Salima and Mulanje district hospitals using a pilot trial, with a multiple-baseline design. To achieve this goal, the investigators will enroll 200 depressed adults living with HIV in the trial, survey patient participants at enrollment, 3-months and 6-months, abstract clinical data related to HIV and depression care, track engagement in the stigma reduction intervention, assess intervention sessions for fidelity to the intervention protocol and conduct qualitative interviews with a sub-set of patients who received the stigma-reduction intervention (n=20) and healthcare providers including HTC counselors (N=4), ART providers (N=10), Friendship Bench counselors (N=6), and counselors (n=4) who deliver the stigma-reduction intervention.

This innovative research will a) address HIV, MI and intersectional stigma while leveraging existing mental health services for people living with HIV, b) lay the ground-work for a multi-level stigma-reduction intervention package, and c) yield detailed insights into barriers and facilitators of implementing stigma-reduction interventions in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV and receiving ART at Salima or Mulanje District Hospital
* Adult (18+ years)
* Elevated depressive symptoms (PHQ-9 Score ≥5)

Exclusion Criteria:

* Pregnant women
* Severe mental or physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the HIV-Mental Illness Stigma Reduction Intervention | Upon the completion of intervention delivery for all patients (assessed up to 6 months)
  The investigators will measure feasibility by conducting qualitative interviews (guided by Proctor's Outcomes for Implementation Research) with providers and counselors who deliver the stigma-reduction intervention. This interview will consist of 12 open-ended questions (with subparts) meant to elicit a response from providers about their perceived changes in their patients' attitudes/well-being, their personal comfort level with delivering the intervention and competency, their training satisfaction, their recommendations for improving the intervention, and their perceived barriers and facilitators to implementation of the intervention.
Patient Acceptability of the HIV-Mental Illness Stigma Reduction Intervention | After completion of all intervention sessions, an average of 6 months
  The investigators will conduct audio-recorded semi-structured qualitative interviews with patients enrolled in the study who initiated depression treatment during the implementation phase. The investigators will use interview guides (using guidance from Proctor's Outcomes for Implementation Research) to conduct qualitative interviews with patients. The interviews will consist of 11 open-ended questions (with subparts) which are designed to elicit a response from the patient about their perceived acceptability of the intervention. This includes how helpful patients believed the intervention was in improving their mental health and feelings of stigma, barriers and facilitators to engagement in the intervention, and perceived areas of improvement and harm of the intervention.
Patient Acceptability of the HIV-Mental Illness Stigma Reduction Intervention | After completion of each intervention session
  The investigators will measure acceptability of the intervention through a quantitative questionnaire, the Client Satisfaction Questionnaire-8. Each of the 8 questions are scored from 1-4 with higher ratings indicating greater satisfaction with the intervention.
Provider Acceptability of the HIV-Mental Illness Stigma Reduction Intervention | Upon intervention delivery completion for all patients (assessed up to 6 months)
  The investigators will use interview guides (using guidance from Proctor's Outcomes for Implementation Research) to conduct qualitative interviews with counselors and providers who deliver the stigma-reduction intervention to assess acceptability to providers. This interview will consist of 12 open-ended questions meant to elicit a response from providers about their perceived changes in their patients' attitudes/well-being, their personal comfort level with delivering the intervention and competency, their training satisfaction, their recommendations for improving the intervention, and their perceived barriers and facilitators to implementation of the intervention.
Fidelity of the Content of the HIV-Mental Illness Stigma Reduction Intervention | Through study completion, an average of 6 months
  The investigators will monitor fidelity in the content of the intervention protocol by assessing the extent to which providers correctly deliver depression treatment and stigma-reduction intervention by reviewing audio-recorded intervention sessions with patients using a fidelity checklist.
Fidelity of the Coverage of the HIV-Mental Illness Stigma Reduction Intervention | Through study completion, an average of 6 months
  The investigators will monitor fidelity in the coverage of the intervention protocol using clinical and program data to measure the percentage of patients who receive the correct depression treatment and the stigma-reduction intervention.
Fidelity of the Frequency of the HIV-Mental Illness Stigma Reduction Intervention | Through study completion, an average of 6 months
  The investigators will monitor fidelity in the frequency of the intervention protocol using clinical and program data to measure the number of completed depression treatment appointments and stigma-reduction intervention sessions, as well as the number of patients who complete the depression treatment and stigma-reduction intervention.
Fidelity of the Duration of the HIV-Mental Illness Stigma Reduction Intervention | Through study completion, an average of 6 months
  The investigators will monitor fidelity in the duration of the intervention protocol using clinical and program data to measure the number of depression treatment and stigma-reduction intervention sessions patients receive over their first six months in HIV care and the attendance of at least 75% of scheduled depression treatment appointments and stigma-reduction intervention sessions (y/n) over the first six months in HIV care.
Preliminary Effectiveness of The HIV-Mental Illness Stigma Reduction Intervention to Reduce Stigma | At enrollment, 3-months post enrollment, and 6-months post enrollment
  Internalized AIDS-Related Stigma Scale will be used to assess patient's level of internalized HIV stigma. Patients rate their agreement of 6 statements. Items are scored with a 0 for disagree or 1 for agree. A higher total scores indicate greater internalized stigma.
Preliminary Effectiveness of The HIV-Mental Illness Stigma Reduction Intervention to Reduce Stigma | At enrollment, 3-months post enrollment, and 6-months post enrollment
  The Adapted Internalized Stigma of Mental Illness Scale will be used to assess patient's level of internalized HIV stigma. The Adapted Internalized Stigma of Mental Illness Scale measures patient's internalized stigma with regard to their mental health. Patients rate their agreement with 29 statements across five subscales: alienation, stereotype endorsement, perceived discrimination, social withdrawal, and stigma resistance. The scale for scoring items indicates a 0 for "strongly disagree" to a 4 for "strongly agree". A higher total scores indicate greater internalized stigma.
Preliminary Effectiveness of The HIV-Mental Illness Stigma Reduction Intervention to Address Depression | At enrollment, 3-months post enrollment, and 6-months post enrollment
  The investigators will utilize the Patient Health Questionnaire (PHQ-9), completed by providers, to measure patients' severity of depression. Patients will indicate how often they experienced 9 depression symptoms in the last 2 weeks. The scale for scoring items indicates a 0 for "not at all" and a 3 for "nearly every day". Higher total scores indicate greater depression severity. Scores of 5 or more are indicative of mild to severe depression.
Preliminary Effectiveness of The HIV-Mental Illness Stigma Reduction Intervention to Improve HIV Care Engagement | Through study completion, an average of 6 months
  Clinical data related to antiretroviral therapy appointment attendance will be abstracted.
Preliminary Effectiveness of The HIV-Mental Illness Stigma Reduction Intervention to Improve HIV Care Engagement | Through study completion, an average of 6 months
  Clinical data related to antiretroviral therapy pill counts will be abstracted.

CONTACTS AND LOCATIONS:
Locations (2):
- Malawi (2):
  - Mulanje District Hospital, Mulanje
  - Salima District Hospital, Salima